CLINICAL TRIAL: NCT05664932
Title: Evaluate the Immunogenicity and Safety of a Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001 as Booster Vaccination in Adults 18 Years of Age or Above Who Have Completed Two-dose or Three-dose Inactivated COVID-19 Vaccine
Brief Title: Immunogenicity and Safety of COVID-19 Vaccine as a Booster Vaccination in Population Aged 18 Years and Above
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangzhou Patronus Biotech Co., Ltd. (Industry)
Collaborators: Yantai Patronus Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LYB001/CT-CHN-301
Record Dates: First submitted 2022-12-23; First posted 2022-12-27 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — ZF2001 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LYB001 Booster Group (Experimental): Subjects 18 years of age or older who has completed two or three-dose inactivated COVID-19 will receive 30μg LYB001 at day 0 as a booster vaccination.
  Interventions: Biological: Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001
- ZF2001 Booster Group (Active Comparator): Subjects 18 years of age or older who has completed two or three-dose inactivated COVID-19 will receive ZF2001 at day 0 as a booster vaccination.
  Interventions: Biological: ZF2001

INTERVENTIONS:
Biological: Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001 — Intramuscular injection of Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001 in the deltoid muscle of the upper arm at day 0. The inoculation dose is 0.5 mL.
  Arms: LYB001 Booster Group
Biological: ZF2001 — Intramuscular injection of ZF2001 in the deltoid muscle of the upper arm at day 0. The inoculation dose is 0.5 mL.
  Arms: ZF2001 Booster Group

SUMMARY:
A total of 1200 people aged 18 years and older who have completed two or three-dose inactivated COVID-19 vaccine for 6-18 months will be recruited in this study. Subjects will be received 1 dose at day 0 as a booster vaccination.Immunogenicity and safety of Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001 will be evaluated.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, positive control design and 1200 subjects are randomly assigned to LYB001 and positive control groups in a 1:1 ratio to evaluate the safety and immunogenicity as a booster vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 years and older, including both males and females;
* Subjects who agree to participate in this clinical trial voluntarily and sign the informed consent form, are capable of providing valid identification, understanding and complying with the requirements of the clinical protocol.
* Subjects who have been vaccinated with two-dose or three-dose inactivated COVID-19 vaccine for 6-18 months .
* For female participants of childbearing potential, effective contraception measures should be used within 2 weeks prior to participation in this study and the results of pregnancy test is required to be negative. Participants should voluntarily agree to use effective contraceptive measures from the time of signing the informed consent form to the end of the study (effective contraceptive measures including oral contraceptives (excluding emergency contraceptives), injectable or implantable contraceptives, sustained-release topical contraceptives, hormonal patches, intrauterine device, sterilization, abstinence, condoms (for males), diaphragms, cervical caps, etc.).

Exclusion Criteria:

* Receipt of any COVID-19 prophylactic medication other than inactivated COVID-19 vaccine (e.g., receipt history of any approved or under developing COVID-19 vaccines, or other COVID-19 prophylactic medication, etc.), or previous vaccination history other than two- or three-dose inactivated COVID-19 vaccination;
* Systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg or axillary body temperature ≥ 37.3°C prior to enrolment;
* Known allergy, or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients;
* History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS);
* History of COVID-19, or close contact with a confirmed/suspected COVID-19 patient or positive results for SARS-CoV-2 nucleic acid ;
* Receipt of any live attenuated vaccine within 28 days prior to vaccination, and other vaccines such as subunit and inactivated vaccine within 14 days prior to vaccination;
* Receipt of blood or blood-related products, including immunoglobulins, monoclonal antibodies, within 3 months prior to vaccination; or any planned use during the study period.
* Subjects with the following diseases:

  1. Any acute diseases or acute attacks of chronic diseases within 7 days prior to enrolment；
  2. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.；
  3. Congenital or acquired immunodeficiency or autoimmune disease, or long-term receipt (>14 consecutive days) of glucocorticoid (reference value for dose: ≥20 mg/day prednisone or equivalent) or other immunosuppressive agents within the past 6 months, with exception of inhaled or topical steroids, or short-term use (≤14 consecutive days) of oral corticosteroids；
  4. Currently suffering from or diagnosed with infectious diseases, such as hepatitis B, hepatitis C, syphilis, AIDS etc.；
  5. History or family history of neurological disorders (convulsions, epilepsy, encephalopathy, etc.) or psychiatric disorders；
  6. Asplenia, or functional asplenia；
  7. Presence of severe, uncontrollable or hospitalized cardiovascular diseases, endocrine diseases, blood and lymphatic diseases, immune diseases, liver and kidney diseases, respiratory diseases, metabolic and skeletal diseases, or malignant tumors;
  8. Contraindications to IM injections and blood draws, such as coagulation disorders, thrombotic or bleeding disorders, or conditions that needs continuous anticoagulant usage.
* Drug or alcohol abuse (alcohol intake ≥ 14 units per week) which in the investigator's opinion would compromise the participant's safety or compliance with the study procedures;
* Pregnant or lactating females;
* Having participated or participating in COVID-19 related clinical trials, and those participating or planning to participate in other clinical trials during the study period;
* Presence of any underlying disease or condition which, in the opinion of the investigator, may place the subject at unacceptable risk, is unable to meet the requirements of the protocol, or interfere with the assessment of vaccine response

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Geometric neutralizing titers (GMT) of neutralizing antibody against variants of concern(VOCs) | Day 14 after booster vaccination
  Geometric neutralizing titers (GMT) of neutralizing antibody against variants of concern(VOCs) at day 14 after booster vaccination in cohort 1.

SECONDARY OUTCOMES:
Geometric mean fold rise(GMFR) of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs) | Day 14 ,day 28 ,month 6 after vaccination
  Geometric mean fold rise(GMFR) of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs) at day 14, day 28, month 6 after booster vaccination in cohort 1.
Seroconversion rate of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs). | Day 14 ,day 28 ,month 6 after vaccination
  Seroconversion rate of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs) at day 14, day 28, month 6 after booster vaccination in cohort 1.
Geometric neutralizing titers (GMT) of neutralizing antibody against SARS-CoV-2 wild strain | Day 14 ,day 28 ,month 6 after vaccination
  Geometric neutralizing titers (GMT) of neutralizing antibody against SARS-CoV-2 wild strain at day 14, day 28, month 6 after booster vaccination in cohort 1.
GMT of binding antibody against SARS-CoV-2 S protein | Day 14 ,day 28 ,month 6 after vaccination
  GMT of binding antibody against SARS-CoV-2 S protein at day 14, day 28, month 6 after booster vaccination in cohort 1.
Geometric mean fold rise(GMFR) of binding antibody against SARS-CoV-2 S protein | Day 14 ,day 28 ,month 6 after vaccination
  Geometric mean fold rise(GMFR) of binding antibody against SARS-CoV-2 S protein at day 14, day 28, month 6 after booster vaccination in cohort 1.
Seroconversion rate of binding antibody against SARS-CoV-2 S protein | Day 14 ,day 28 ,month 6 after vaccination
  Seroconversion rate of binding antibody against SARS-CoV-2 S protein at day 14, day 28, month 6 after booster vaccination in cohort 1.
The occurrence of adverse events | 30 mins,7 days and 28 days after vaccination
  The occurrence of adverse events within 30 mins,7 days and 28 days after each vaccinatio
The occurrence rate of serious adverse events (SAEs) and adverse events of special interest (AESIs) | Day 0 to 12 months after vaccination
  The occurrence rate of serious adverse events (SAEs) and adverse events of special interest (AESIs) within 12 months after vaccination（28 days after vaccination for positive control group）

CONTACTS AND LOCATIONS:
Overall Officials: Xianfeng Zhang, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Hubei Provincial Center for Disease Control and Prevention, Wuhan, Hubei, China

REFERENCES:
- [Derived] Yang BF, Jin J, He XR, Yang ZH, Qian X, Tong YQ, Ke CX, Li ZH, Li ZX, Zhong LF, Gan ZH, Zhang XF, Zeng Y. Immunogenicity and safety of SARS-CoV-2 recombinant protein vaccine (CHO cell) LYB001 as a heterologous booster following two- or three-dose inactivated COVID-19 vaccine in adults aged >/=18 years: interim results of a randomized, active-controlled, double-blinded, phase 3 trial. Expert Rev Vaccines. 2025 Dec;24(1):81-90. doi: 10.1080/14760584.2024.2446288. Epub 2025 Jan 5. PMID 39720838